CLINICAL TRIAL: NCT05934071
Title: Evaluation of the Effects of the Sodium-glucose Cotransporter 2 Inhibitors+Sacubitril/Valsartan Combined Therapy in Patients With HFrEF: an Echocardiographic Study.
Brief Title: Effects of the Sodium-glucose Cotransporter 2 Inhibitors+Sacubitril/Valsartan Therapy in Patients With HFrEF.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5428
Record Dates: First submitted 2023-03-03; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure; Ventricular Remodeling; Ventricular Dysfunction
MeSH Terms: conditions — Heart Failure; Ventricular Remodeling; Ventricular Dysfunction | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: None Retained — blood sample
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients affected by HFrEF on ARNI: patients affected by HFrEF in optimized medical therapy including ARNI, eligible for glyphozine
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — optimization of the medical therapy for heart failure with reduced ejection fraction with SGLT2 inhibitor, according to clinical guidelines
  Other Names: Dapaglifozin, Empaglifozin

SUMMARY:
The goal of this observational study is to investigate the effects of combination therapy with ARNI and inhibitors of SGLT2 in patients affected by HFrEF.

The main questions it aims to answer are:

* What is the medium-long term impact of the ARNI + glyphozine combination therapy in terms of ventricular remodeling studied by speckle tracking echocardiography (GLS%) and by variation of volumetric indices and contractile function (LVEDV, LVEDD, FE%)?
* What is the medium-long term impact of the ARNI + glyphozine combination therapy in terms of variation of laboratory data indicative of heart failure (NT-pro-BNP)?
* What is the medium-long term impact of the ARNI + glyphozine combination therapy in terms of major cardiovascular events (MACVE)?
* What are the echocardiographic and laboratory parameters predictors of medium-long term major cardiovascular events (MACVE) and ventricular remodeling? Participants will undergo, at the time of enrollment and after approximately 3 and 12 months from the introduction of SGLT-2 inhibitor therapy, at clinical, echocardiographic and biohumoral investigations.

DETAILED DESCRIPTION:
According to the 2021 ESC guidelines for heart failure, iSGLT2 has become the cornerstone of the treatment of heart failure with reduced ejection (HFrEF) fraction, with a class of recommendation IA (1).

However, the mechanisms of action of iSGLT2 remain still little known. In particular, if the combined therapy with ARNI and iSGLT2 may have an effect in terms of left ventricular remodeling evaluated by speckle tracking echocardiography (GLS%) in patients with HFrEF at a medium-long term (3-12 months) is still to be defined (primary objective).

Furthermore, our study will aim to evaluate the clinical and echocardiographic impact of the combined therapy with ARNI + iSGLT2 in terms of left ventricular remodeling evaluated through volumetric and contractile function indices (LVEDV, LVEDD, FE%) and in terms of variation of laboratory data suggestive of decompensated heart failure (NT-pro-BNP) in patients with HFrEF at a medium-long term follow-up (3-12 months) (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* HFrEF on ARNI
* Ability to express written informed consent to participate in the study

Exclusion Criteria:

* Contraindication to glyphozine therapy (i.e., severe renal insufficiency with filtration estimated glomerular <30ml/min/m2 or history of recurrent urinary tract infections);
* Comorbidities with expected survival of less than 1 year;
* Limited or legal inability to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by HFrEF on ARNI, eligible for glyphozine
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ventricular remodeling studied by speckle tracking echocardiography | 3-12 months
  Evaluation of the medium-long term impact of the ARNI + glyphozine combination therapy in terms of ventricular remodeling studied through speckle tracking echocardiography and evaluated in terms of global longitudinal strain values (GLS%)

SECONDARY OUTCOMES:
variation of volumetric indices and contractile function | 3-12 months
  Evaluation of the medium-long term impact of the ARNI + glyphozine combination therapy in terms of ventricular remodeling studied through echocardiography and evaluated as LV volumes (end diastolic volumes-ml/m2 and and systolic volumes ml/m2) and LV function (left ventricular ejection fraction-%) indices
variation of laboratory data indicative of heart failure (NT-pro-BNP) | 3-12 months
  Evaluation of the medium-long term impact of the ARNI + glyphozine combination therapy in terms of variation of laboratory data indicative of heart failure (N-terminal pro B type natriuretic peptide-pg/mL)
major cardiovascular events (MACVE) | 3-12 months
  Evaluation of the medium-long term impact of the ARNI + glyphozine combination therapy in terms of major adverse cardiovascular events (composite endpoint of all-cause mortality, non-fatal myocardial infarction, non-fatal stroke)
echocardiographic and laboratory parameters predictors of medium-long term major cardiovascular events (MACVE) and ventricular remodeling | 3-12 months
  Identification of the echocardiographic and laboratory parameters predictors of medium-long term major cardiovascular events (MACVE) and ventricular remodeling in terms of variation of LV volumes (end diastolic volumes-ml/m2 and and systolic volumes ml/m2) and LV function (left ventricular ejection fraction-%) indices

CONTACTS AND LOCATIONS:
Overall Officials: NADIA ASPROMONTE, Prof., Principal Investigator — Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy.
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCSS, Roma, RM, Italy